CLINICAL TRIAL: NCT02920619
Title: The ULTRA Study: Cross-Comparison of Muscle Composition Measures in Multiple Ultrasound Systems
Brief Title: The ULTRA Study: Cross-Comparison of Ultrasound Systems
Acronym: ULTRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Harris-Love, Associate Director, CRC Human Performance Research Unit, Washington D.C. Veterans Affairs Medical Center
Other Study IDs: MIRB01803
Record Dates: First submitted 2016-09-24; First posted 2016-09-30 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Healthy
Keywords: ultrasound; muscle
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Ultrasound — Imaging of the rectus femoris, lower-trapezius, brachioradialis, tibialis anterior, middle deltoid, and pectoralis major will be conducted in Veteran participants during a single visit to the Washington D.C. Veterans Affairs Medical Center. Imaging will be conducted by investigators experienced with quantitative ultrasound using diagnostic musculoskeletal B-mode ultrasound with a 10 Mhz linear transducer.

SUMMARY:
The purpose of this study is to develop computational methods for cross-comparison of muscle composition measurements in three laboratory ultrasound systems.

DETAILED DESCRIPTION:
The purpose of this study is to develop computational methods for cross-comparison of muscle composition measurements in three laboratory ultrasound systems. We propose a cross-sectional study to obtain ultrasound images of selected muscles in Veteran participants. These data will be used to develop conversion models for each system. Evaluation of neuromuscular symptoms such as muscle weakness and fatigue is crucial to improving quality of life among Veterans. These symptoms may be related to progressive changes in muscle tissue composition, including increased intramuscular fat and atrophy. Quantitative musculoskeletal ultrasound is a diagnostic imaging application used to characterize muscle tissue composition. Despite its non-invasiveness and relative low cost, quantitative musculoskeletal ultrasound has not been widely adopted by the medical community due in part to technical barriers that impede generalization of measurements across ultrasound systems. Unfortunately, few techniques have been proposed to reliably compare system measurements. Development of new cross-comparison methods could expand quantitative musculoskeletal ultrasound applications and improve neuromuscular symptoms diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female Veteran who receives medical care at the Washington DC VA Medical Center
* Ages 20-85

Exclusion Criteria:

* Limb amputation (upper or lower extremity)
* Lower extremity joint replacement
* Severe cognitive impairment
* Edema
* Inability to read, speak, or understand English

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Thirty adult Veterans (20-85 years) will be recruited for the study from the DC VAMC.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-09 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Echogenicity | 1 day
  Echogenicity values (i.e., image brightness) obtained from the ultrasound scans (units: grayscale levels, 0-255)

SECONDARY OUTCOMES:
Muscle thickness | 1 day
  Morphometry values (units: cm) obtained from the ultrasound scans using digital calipers.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Harris-Love, D.Sc., Principal Investigator — Washington DC VA Medical Center
Locations (1):
- Washington DC VA Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harris-Love MO, Seamon BA, Teixeira C, Ismail C. Ultrasound estimates of muscle quality in older adults: reliability and comparison of Photoshop and ImageJ for the grayscale analysis of muscle echogenicity. PeerJ. 2016 Feb 22;4:e1721. doi: 10.7717/peerj.1721. eCollection 2016. PMID 26925339